CLINICAL TRIAL: NCT02900898
Title: Effect of a Dynamic Exercise Program in Combination With a Mediterranean Diet on Body Composition, Strength, Inflammatory Markers, Joint Mobility and Disease Activity in Women With Rheumatoid Arthritis
Brief Title: Exercise and Mediterranean Diet on Body Composition, Disease Activity and Inflammatory Markers in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LILIA CASTILLO MARTINEz (Other)
Responsible Party: Sponsor-Investigator, LILIA CASTILLO MARTINEz, Medical Research Scientist, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Organization: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIC004
Record Dates: First submitted 2016-08-24; First posted 2016-09-14 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Arthritis, Rheumatoid; Dietary Modifications; Motor Activity; Body Composition, Beneficial; Physical Activity; Inflammation
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity; Glucocorticoid Receptor Deficiency; Inflammation | interventions — Diet, Mediterranean; Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dynamic exercise and Mediterranean diet (Experimental): DE: divided in stretch: arms, hands, legs, knees, for 20 seconds (s), resting 5, warming and flexion: making small circles forward and backward for 20 s, resting 5, DE: resistance (contraction, twisting) using therapeutic leagues with 20 repetitions, resting 10 s. Aerobic part will perform in a treadmill by 20 minutes (monitoring blood pressure and heart rate) and relaxation: involved the "stretching" part.
  MD: Individualized diet (energy expenditure) according to age, ideal weight and height. Distribution of macronutrients will be 50% carbohydrates, 30% lipids and 20% of proteins. This diet is according to the Mediterranean diet patterns and consist in five meals: breakfast, snack, principal meal, snack and dinner. All recommended meals include type of food and method of preparation.
  Interventions: Other: Dynamic exercise and Mediterranean diet
- Dynamic exercise (Experimental): DE: divided in stretch: arms, hands, legs, knees, for 20 seconds (s), resting 5, warming and flexion: making small circles forward and backward for 20 s, resting 5, DE: resistance (contraction, twisting) using therapeutic leagues with 20 repetitions, resting 10 s. Aerobic part will perform in a treadmill by 20 minutes (monitoring blood pressure and heart rate) and relaxation: involved the "stretching" part.
  Interventions: Other: Dynamic exercise
- Mediterranean diet (Experimental): MD: Individualized diet (energy expenditure) according to age, ideal weight and height. Distribution of macronutrients will be 50% carbohydrates, 30% lipids and 20% of proteins. This diet is according to the Mediterranean diet patterns and consist in five meals: breakfast, snack, principal meal, snack and dinner. All recommended meals include type of food and method of preparation.
  Interventions: Other: Mediterranean diet
- Control (Active Comparator): This group will not carry out interventions.
  Interventions: Other: Control

INTERVENTIONS:
Other: Dynamic exercise and Mediterranean diet — DE, MD
  Other Names: Diet and physical treatment
  Arms: Dynamic exercise and Mediterranean diet
Other: Dynamic exercise — DE
  Other Names: Physical treatment
  Arms: Dynamic exercise
Other: Mediterranean diet — MD
  Other Names: Diet treatment
  Arms: Mediterranean diet
Other: Control — Control
  Arms: Control

SUMMARY:
Rheumatoid arthritis (RA) is a chronic autoimmune disease with metabolic alterations due mainly by the liberation of catabolic cytokines leading to changes in body composition as rheumatoid cachexia. Dynamic exercise (DE) has demonstrated to improve muscular, strength and joint function as well as inflammatory process. Also, a diet focused on the consumption of certain fatty acids like the Mediterranean is recommended to reduce inflammation. The aim of this study is to assess the effect of a dynamic exercise program in combination with a Mediterranean diet in strength, joint mobility and disease activity in women with RA.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic autoimmune disease characterized by inflammation, joint pain, destruction of the synovial membranes and metabolic alterations due mainly by the liberation of tumor necrosis factor alpha and interleukin-1 beta mainly and leading to changes in body composition as rheumatoid cachexia, which is characterized by involuntary loss of muscular mass with or without loss of body weight and with or without gain of fat mass and therefore reducing physical activity and affecting nutrition. Alternative therapies that could improve these metabolical changes are "Dynamic exercise" (DE) which has demonstrated to improve muscular function and muscular strength, as well as joint mobility and joint inflammatory markers without negative effects on RA. Also, "Mediterranean diet" (MD) which is recommended to reduce inflammation by the high intake of monounsaturated and polyunsaturated and low in saturated fats. Previous studies report the benefits of nutritional interventions but in the majority of the cases therapies are based on specific foods and not in the form of diet. Likewise, physical interventions are different regarding in time and type of movement. However both interventions have shown ambiguous findings in terms of body composition (mainly) and which prevents drawing conclusions and generate recommendations on the implementation of these therapies (in combination). As far as the investigators know, no studies evaluating the effect of a diet and exercise combined. Thus the aim of this study is to assess the effect of DE program in combination with a MD on body composition, strength, joint mobility and disease activity in women with RA.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Women (nonpregnant).
* Patients with confirmed RA and functional classification I - III.
* Patients who voluntarily accept previously signed informed consent

Exclusion Criteria:

* Patients participating in other investigations.
* Patients with chronic renal failure, cancer, HIV, heart failure.
* Patients with inability to perform physical exercises.
* Patients who make a structured exercise plan (rehabilitation) at the time of inclusion in the study.
* Patients with systemic lupus erythematosus, psoriatic arthritis, gout, fibromyalgia, scleroderma, Sjögren's syndrome or some other autoimmune pathology.
* Patients with functional class IV.
* Patients with partial or total joint replacement.
* Patients who are taking any dietary supplement at the time of inclusion in the study.
* Patients who are treated with biological drugs.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in body composition by bioelectric impedance analysis at 24 weeks after dynamic exercise program in conjunction with a diet based on the Mediterranean pattern | 24 weeks
  Change in resistance, reactance, phase angle. Impedance vector analysis

SECONDARY OUTCOMES:
Change from baseline in muscular strength | 24 weeks
  Change from baseline in muscular strength by hand dynamometry at 24 weeks after dynamic exercise program in conjunction with a diet based on the Mediterranean pattern
Change from baseline in inflammatory cytokines and chemokines by spectrophotometry | 24 weeks
  Change from baseline in inflammatory cytokines and chemokines by spectrophotometry assay ELISA at 24 weeks after dynamic exercise program in conjunction with a diet based on the Mediterranean pattern
Change from baseline in joint mobility by goniometry | 24 weeks
  Change from baseline in joint mobility by goniometry at 24 weeks after dynamic exercise program in conjunction with a diet based on the Mediterranean pattern
Change from baseline in disease activity by DAS28 | 24 weeks
  Change from baseline in disease activity by DAS28 at 24 weeks after dynamic exercise program in conjunction with a diet based on the Mediterranean pattern
Change from baseline in physical capacity by 6 minute walk test | 24 weeks
  Change from baseline in physical capacity by 6 minute walk test at 24 weeks after dynamic exercise program in conjunction with a diet based on the Mediterranean pattern

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Pineda Juárez, PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Lilia Castillo Martínez, PhD, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Mariel Lozada Mellado, BSc, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Midori Ogata Medel, BSc, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Rocío Cervantes Gaytán, BSc, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Andrea Hinojosa Azaola, MD, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Jorge Alcocer Varela, MD, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Luis Llorente Peters, MD, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Arturo Orea Tejeda, MD, Study Director — Instituto Nacional de Enfermedades Respiratorias Ismael Cosío Villegas
Locations (1):
- Juan Antonio Pineda Juárez, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ogata-Medel M, Llorente L, Hinojosa-Azaola A, Lozada-Mellado M, Pineda-Juarez JA, Rocha-Gonzalez HI, Castillo-Martinez L. Cachexia measured by bioelectrical impedance vector analysis and risk of infection in women with rheumatoid arthritis. Clin Rheumatol. 2023 Feb;42(2):391-397. doi: 10.1007/s10067-022-06431-5. Epub 2022 Nov 14. PMID 36372851
- [Derived] Lozada-Mellado M, Llorente L, Hinojosa-Azaola A, Garcia-Morales JM, Ogata-Medel M, Alcocer-Varela J, Pineda-Juarez JA, Castillo-Martinez L. Comparison of the Impacts of a Dynamic Exercise Program vs. a Mediterranean Diet on Serum Cytokine Concentrations in Women With Rheumatoid Arthritis. A Secondary Analysis of a Randomized Clinical Trial. Front Nutr. 2022 Apr 25;9:834824. doi: 10.3389/fnut.2022.834824. eCollection 2022. PMID 35548581